CLINICAL TRIAL: NCT05776368
Title: Links Between Motor Abilities and Language Ability Deficits in Patients With Post-stroke Aphasia
Acronym: MOTOLANG-AVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL22_0472; 2022-A01229-34 (Other: ID-RCB)
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Aphasia
Keywords: stroke; aphasia; rehabilitation; tool use; Broca's area; basal ganglia; healthy volunteer; language and motor abilities
MeSH Terms: conditions — Stroke; Aphasia; Language | interventions — Mastectomy, Segmental; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Sub-study E1, arm 1, patients and tool motor training (Experimental): patients undergo a 30 minutes tool motor training and two linguistic tasks (one before and one after).
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: Motor training with a tool; Other: linguistic tasks
- Sub-study E1, arm 2, patients and hand motor training (Experimental): patients undergo a 30 minutes hand motor training and two linguistic tasks (one before and one after).
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: Motor training with a hand; Other: linguistic tasks
- Sub-study E1, arm 3, patients and no motor training (control group) (Experimental): patients only undergo two linguistic tasks separated by a 30-minutes break (without motor activity (control group)).
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: linguistic tasks
- Sub-study E1, arm 4, healthy volunteers and tool motor training (Experimental): healthy volunteers undergo a 30 minutes tool motor training and two linguistic tasks (one before and one after).
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: Motor training with a tool; Other: linguistic tasks
- Sub-study E1, arm 5, healthy volunteers and hand motor training (Experimental): healthy volunteers undergo a 30 minutes hand motor training and two linguistic tasks (one before and one after).
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: Motor training with a hand; Other: linguistic tasks
- Sub-study E1, arm 6, healthy volunteers and no motor training (control group) (Experimental): healthy volunteers only undergo two linguistic tasks separated by a 30-minutes break (without motor activity (control group)).
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: linguistic tasks
- Sub-study E2, arm 1, single case design (Experimental): patients undergo 4 weeks of tool motor training according to an on/off design.
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: on/off effect of tool motor training; Other: linguistic tasks
- Sub-study E3, arm 1, patients and 4 week experimental sensorimotor protocol (Experimental): patients undergo 4 weeks of tool motor training
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: Motor training with a tool; Other: linguistic tasks
- Sub-study E3, arm 2, control group of patients (Experimental): aphasic patients receiving the standard treatment as a control group
  Interventions: Other: Syntactic comprehension battery (BCS); Other: Montreal Cognitive Assessment (MOCA); Other: Purdue Pegboard Test; Other: The Box and Block Test (BBT); Other: linguistic tasks

INTERVENTIONS:
Other: Syntactic comprehension battery (BCS) — The BCS is a battery for assessing syntactic skills. In this study, only one part of the BCS will be performed, namely task C2.
  It consists in assessing the ability to assign thematic roles. To do this, the participant selects the image corresponding to the sentence he/she hears on a board of 2 images.
  Task C2 consists of 50 tests of 2 images. A total score is given out of 50 points. The higher the score, the more successful the test.
Other: Montreal Cognitive Assessment (MOCA) — The MOCA is a short 30-question test that assesses several cognitive domains and allows for early detection of cognitive disorders. The MOCA test takes about 10-15 minutes to administer and consists of several sections, the first of which is an assessment of orientation in time and space. Then there are tasks that assess memory, concentration and reasoning ability, as well as language and visuospatial ability tasks.
  The MOCA score can range from 0 to 30 points, with a score of 26 points or more considered normal.
Other: Purdue Pegboard Test — The Purdue Pegboard Test is a test of fine motor skills and hand-eye coordination. The test consists of a perforated board with holes into which participants must insert pegs or counters.
  The assessment consists of four subtests, each repeated 3 times:
  * Right hand (30 seconds): The total number of pins placed in the right column with the right hand in 30 seconds.
  * Left hand (30 seconds): The total number of rods placed in the left column with the left hand in 30 seconds.
  * Two hands (30 seconds): The total number of pairs of rods placed in both columns using both hands simultaneously, in 30 seconds.
  * Assembly (60 seconds): The total number of rods, washers and clamps assembled in the allotted time, using both hands.
Other: The Box and Block Test (BBT) — The Box and Block Test (BBT) is a standardised test of manual dexterity used to assess motor function and hand-eye coordination in people of all ages.
  The subject must move, one by one, a maximum number of cubes from one compartment of the box to another of equal size for 60 seconds. He starts with the healthy upper limb or, if not, with the dominant side. A 15 second trial period is allowed at the beginning of each side.
Other: Motor training with a tool — The patient will do around 30 minutes of motor training with a tool (pliers). They have to put most pieces as possible in the board with the pliers. Patients hold the pliers with the right hand (dominant hand) or with the left one if not possible (motor disorder).
  For E1 Arm1 and E1 Arm 4: the participant will do the motor training with a tool one time in this study.
  For E3 Arm 1: the participant will do the motor training with a tool During 4 weeks (3 to 5 training sessions of 30 minutes)
  Arms: Sub-study E1, arm 1, patients and tool motor training; Sub-study E1, arm 4, healthy volunteers and tool motor training; Sub-study E3, arm 1, patients and 4 week experimental sensorimotor protocol
Other: Motor training with a hand — The patient will do around 30 minutes of motor training with the hand. They have to put most pieces as possible in the board with the right hand (dominant hand) or with the left one if not possible (motor disorder).
  Arms: Sub-study E1, arm 2, patients and hand motor training; Sub-study E1, arm 5, healthy volunteers and hand motor training
Other: on/off effect of tool motor training — During 4 weeks, patients switch between tool training weeks ("on") and control weeks ("off") during which they don't practice motor training.
  During "on" weeks they do 3 to 5 tool motor training sessions of 30 minutes. They use pliers with the right hand (dominant hand) or with the left one if not possible (motor disorder) and have to put most pieces as possible in the board.
  During "off" weeks they do 3 to 5 control sessions where they only do the two linguistic tasks separated between a 30-minutes break.
  Arms: Sub-study E2, arm 1, single case design
Other: linguistic tasks — The linguistic tasks consists in the presentation of correct sentences at the center of a computer screen. The sentence can be a coordinated one (" The policeman stopped the woman and asked the question "), or a subject relative (i.e., " The policeman who stopped the woman asked the question "), or an object relative (" The policeman who the woman stopped asked the question "). After the sentence an affirmation test is proposed of the kind " the policeman stopped the woman ", and the participant has to respond ads quick as possible whether it is true or false.

SUMMARY:
Aphasia is a language disorder that affects oral and written expression and/or comprehension. It's one of the most disabling consequence of stroke. Nowadays, aphasia rehabilitation is supported by speech therapists and is based on oral and written language, comprehension and expression. However recent studies have shown links between language and motor function (especially tool use). Two domains that share neural substrates (Broca's area, basal ganglia) and that can influence each other.

The aim of this study is to show that a motor training with a tool (pliers) can improve short-term and long-term language abilities of aphasic patients who had a stroke at least 3 months ago.

The investigators hypothesis is that there is a learning transfer between tool use and language abilities in aphasic patients with an inferior frontal gyrus (IFG) lesion caused by a stroke, thanks to their shared neural resources.

Investigators aim to study long and short-time effects of this tool motor training with three experiments:

* E1 will study short-term effects by estimating pre-post effect of a motor training on language abilities. Investigators will experiment different effectors: tool, hand, none (control group); on patients and healthy volunteers.
* E2 will study long-term effects with multiple single-case experimental designs (SCED). Patients will undergo four weeks of on-off design.
* E3 will study long-term effects by estimating the efficiency of an experimental sensorimotor protocol of four weeks, comparing a group of patients with the experimental sensorimotor protocol to a control group of patients

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Adult male or female aged 18 years and over
* Right-handed
* Having signed an informed and written consent
* Affiliated to a social security scheme
* Have French as their first language

For patients :

* Left inferior frontal gyrus lesion following a stroke
* Stroke more than 3 months old
* Aphasia proven by a pathological score on the A-2 test of the Syntax Comprehension Battery (BCS)

Exclusion Criteria:

For all participants:

* Cognitive abilities that prevent completion of the study tasks (assessed with the MOntreal Cognitive Assesment (MOCA))
* Language skills impaired by other disorders (for example neurodegenerative disease)
* Cognitive impairing treatments (for example psychotropic drugs)
* Neurovisual disorder (hemineglect, unilateral spatial neglect)
* Impairment of both upper limb abilities that prevent motor training (pathological score in the Purdue Pegboard Test and/or Box and Block Test).
* Recurrence of a stroke impacting the reorganisation of neural networks
* Persons deprived of their liberty by a judicial or administrative decision Persons of legal age under a legal protection measure (guardianship, curatorship)
* Pregnant women, women in labour or nursing mothers, confirmed by questioning the participant
* Participation in another study at the same time as this one

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
reaction time | 4 weeks following the inclusion
  This is defined as the time necessary to give a correct answer to the affirmation test. It is calculated at each trial of the syntactic task as the time between the appearance of the affirmation test and the time when a correct answer is provided by the patient. The unit of measure is millisecond. An average is then calculated for each condition (i.e. for each sentence type), at each time point.
sensitivity index | 4 weeks following the inclusion
  The sensitivity index is a measure of the accuracy of response which also takes into account the false alarms. It gives a measure of how the patient can distinguish the signal (correct syntax) from noise (incorrect syntax). It is calculated as the difference between the standardized proportion of correct responses (answer " True " correct) and the standardized proportion of fall alarms (answer " True " incorrect). It is expressed in zed points.

SECONDARY OUTCOMES:
number of inserted pieces | 4 weeks following the inclusion
  The evolution of motor performance is represented by the number of inserted pieces during the nine training blocks of two minutes each.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Equipe ImpAct CRNL, Bron
  - Hôpital neurologique Pierre Wertheimer, Bron
  - Hôpital Henry Gabrielle, Saint-Genis-Laval